CLINICAL TRIAL: NCT02228694
Title: IMPact of a Regulated ADC System On Medication Distribution and Administration VariablEs
Brief Title: The IMPROVE Study-IMPact of a Regulated ADC System
Acronym: IMPROVE
Status: Completed | Type: Observational
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Omnicell (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00004749
Record Dates: First submitted 2014-08-08; First posted 2014-08-29 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Medication Administered in Error; Medication Compliance
Keywords: ADC; Pre installation; Post installation; Safety; Time
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
An automated dispensing cabinet (ADC) is a computerized drug storage device or cabinet designed for hospitals. ADCs allow medications to be stored and dispensed near the point of care while controlling and tracking drug distribution.This study seeks to obtain quantitative measurements of the impact of the regulated ADC System installed in select high volume units throughout the hospital.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the impact of the regulated ADC Systems on the medication administration processes. HackensackUMC is specifically interested in measuring the time to first dose administration from scheduled dosing times of the IV antibiotic piperacillin and tazobactam for injection, USP. and we are interested in assessing a reduction in time from scheduled dosage times of first dose to documented administration after the implementation of the regulated ADC system compared to before.

Timely administration of antibiotics improves morbidity, mortality, and length of hospital stay.Early and effective antibiotic therapy is essential in the management of infection in critical illness. The loading dose is probably the most important dose and is a function of the volume of distribution of the drug and the desired plasma concentration but independent of renal function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects treated at study site in units where regulated ADC System was installed where greater number of medications is administered due to patient volume per nurse assignment or where greater throughput occurs
* Time-sensitive scheduled medications administered on units where administration includes the use of the medication label printer
* Piperacillin and tazobactam for injection, USP (United States Pharmacopeia)
* All IV antibiotics
* Insulin
* Heparin

Exclusion Criteria:

* Medication administration data prior to January 1, 2013;
* Medication administration data after March 31, 2013 through December 31, 2013;
* Medication administration data after March 31, 2014.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Number of Participants by Group
  * Children (Minor Subjects): 0
  * Cognitively Impaired Participants:0
  * Employees and Students: 120
  * Patients: 25238
  * Prisoners: 0
  * Normal Healthy Volunteers: 0
  * Pregnant Women-Human Fetuses: 0
  * Wards: 0
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Medication Administered in Error | six months
  Medication error rates for heparin and insulin pre-install of regulated ADC system compared to post installation. For each drug, heparin and insulin, the number of medication errors will be enumerated based on event type of the voluntary reporting event report data. For each drug, medication error rates will be calculated by dividing the number medication errors by the number of medication orders multiplied by 1,000. Comparison of medication error rates pre-install and post-install will be conducted using simple Poisson regression analysis obtained in, results of which will be expressed as incidence rate ratio (IRR) and 95% confidence intervals (CI).

SECONDARY OUTCOMES:
Timeliness of medication administration | six months
  We are measuring timeliness of medication administration - CMS describes time-critical scheduled medications as those scheduled medications that are identified under the hospital's policies and procedures as time-critical must be administered within thirty minutes before or after their scheduled dosing time, for a total window of 1 hour. First dose IV antibiotics are time-critical. We intend to demonstrate a 10% reduction in time from scheduled dosing times to first dose for the IV piperacillin and tazobactam for injection, USP and for all dose IV antibiotcs post install of the regulated ADC System compared to pre-installation in the medical-surgical, orthopedic, and oncology units.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Douglas, DNP, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical center, Hackensack, New Jersey, United States